CLINICAL TRIAL: NCT02445625
Title: An Interventional Study to Improve Social Attention in Autistic Spectrum Disorder (ASD): A Brain Computer Interface (BCI) Approach
Brief Title: BCI (Brain Computer Interface) Intervention in Autism
Acronym: BCIAUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Responsible Party: Principal Investigator, Miguel Castelo-Branco, MD, PhD, University of Coimbra
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBILI-VB-2015-01
Record Dates: First submitted 2015-04-24; First posted 2015-05-15 (Estimated); Results first posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2018-12

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BCI to train joint attention in ASD (Experimental): We are using Brain Computer Interfaces implemented by EEG in 16 ASD subjects
  Interventions: Device: BCI to train joint attention in ASD

INTERVENTIONS:
Device: BCI to train joint attention in ASD — The intervention comprehends seven BCI sessions spread over four months. The first four sessions are planned to occur weekly, and the rest monthly. In each session, the subject is asked to identify objects of interest based on the gaze direction of an avatar. The subject response is interpreted from the EEG signal (using the P300 component, as established in our previous work).

SUMMARY:
This study aims to demonstrate that improvements in identification of social clues (and improvement of overall social behaviour) in subjects with ASD can be achieved using social games together with a BCI setup.

The primary goal is to ensure increased rate of responses to joint attention cues.

Intervention Type is a Device (brain computer interface using EEG). Structure: (1) initial eligibility screening (within 1 week after admission), (2) pre-intervention (first week of study, baseline outcome measures and additional evaluations), (3) intervention process (16 weeks), (4) post-intervention (outcome measures and additional evaluations), and (5) follow-up (outcome measures at 6 months).

DETAILED DESCRIPTION:
Clinical research has demonstrated that ASD children have deficits in the interpretation of others intentions from gaze-direction or other social attention cues (Baron-Cohen, Baldwin, & Crowson, 1997).

The purpose of the study is to investigate whether a brain computer interface (BCI) using electroencephalographic (EEG) signals can be used to train social cognition skills (in particular interpretation of gaze direction pointing to objects of interest) in ASD patients and whether this improves clinical symptoms.

The intervention comprehends seven BCI sessions spread over four months. The first four sessions are planned to occur weekly, and the rest monthly. In each session, the subject is asked to identify objects of interest based on the gaze direction of an avatar. The subject response is interpreted from the EEG signal (using the P300 component, as established in our previous work).

ELIGIBILITY:
Inclusion Criteria:

* Positive diagnostic results for ASD in:

Autism Diagnostic Interview-Revised; Autism Diagnostic Observation Schedule; The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria.

Exclusion Criteria:

* Global Intelligence Quotient < 80
* Associated medical condition such as epilepsy, neurocutaneous or other genetic syndromes, or other usual comorbidity in ASD samples

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miguel S Castelo-Branco, MD, PhD., Principal Investigator — IBILI - Institute for Biomedical Imaging in Life Sciences

REFERENCES:
- [Background] Baron-Cohen S, Baldwin DA, Crowson M. Do children with autism use the speaker's direction of gaze strategy to crack the code of language? Child Dev. 1997 Feb;68(1):48-57. PMID 9084124
- [Derived] Amaral C, Mouga S, Simoes M, Pereira HC, Bernardino I, Quental H, Playle R, McNamara R, Oliveira G, Castelo-Branco M. A Feasibility Clinical Trial to Improve Social Attention in Autistic Spectrum Disorder (ASD) Using a Brain Computer Interface. Front Neurosci. 2018 Jul 13;12:477. doi: 10.3389/fnins.2018.00477. eCollection 2018. PMID 30061811

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 15 (plus 3 in case of drop outs) participants will be recruited. We expect to recruit one subject each three weeks. We recruited the first participant on the second semester of 2015 and the study last up to 82 weeks (including follow-up).
Groups:
- High Functioning ASD Adolescents and Adults: The eligible patients for the study should be high functioning ASD adolescents and adults.
  These participants should also meet all the following inclusion criteria and none of the exclusion criteria. All queries about patient eligibility should be directed to Susana Mouga before registration. Positive diagnostic results for ASD in:
  * Autism Diagnostic Interview-Revised;
  * Autism Diagnostic Observation Schedule;
  * The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria.
Period: Overall Study
Arm/Group | High Functioning ASD Adolescents and Adults
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | High Functioning ASD Adolescents and Adults
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.333 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Portugal | 15
JAAT_NoFace [Mean (Standard Deviation); unit: Correct Fixations] — Number of fixations on the target object of the joint attention animation of an avatar after the animation starts (e.g. looking at, pointing at) in the Joint-attention assesment task - JAAT_NoFace with no previous fixation on avatar face.. We will use a new task/realistic game that will challenge the detection of initiation of joint attention cues (from avatars - gaze or pointing). The number of correct responses (to particular objects and not to non-object parts of the scene) will be recorded. We will also record incorrect responses to non-pointing body gestures.
  Correct Fixations | 16.33 (9.36)
JAAT_Face [Mean (Standard Deviation); unit: Correct Fixations] — Number of fixations on the target object of the joint attention animation of an avatar after the animation starts (e.g. looking at, pointing at) in the Joint-attention assesment task - JAAT_NoFace with previous fixation on avatar face.. We will use a new task/realistic game that will challenge the detection of initiation of joint attention cues (from avatars - gaze or pointing). The number of correct responses (to particular objects and not to non-object parts of the scene) will be recorded. We will also record incorrect responses to non-pointing body gestures.
  Correct Fixations | 10.67 (9.35)
ATEC - Autism Treatment Evaluation Checklist [Mean (Standard Deviation); unit: score on a scale] — Autism Treatment Evaluation Checklist (ATEC) evaluates the effectiveness of autism treatments - a 1-page form designed to be completed by parents or caretakers. It consists of 4 subtests: I. Speech/Language Communication (14 items, min.0-max.28); II. Sociability (20 items, min.0-max.40); III. Sensory/Cognitive Awareness (18 items, min.0-max.36); and IV. Health/Phys./Behavior (25 items, min.0-max.75). Total score (sum) ranges from min.0-max.179.
  The results reported here correspond to the total ATEC score to be used for comparison at a later date. The lower the score, the fewer the problems.
  score on a scale | 35.57 (12.53)
VABS - Vineland Adaptive Behaviour Scale [Mean (Standard Deviation); unit: units on a scale] — The Vineland Adaptive Behaviour Scale (VABS) is a semi-structured interview designed to assess global adaptive functioning, composed by 3 main domains: Communication COM, Daily Living Skills DLS and Socialization SOC. The Adaptive Behaviour Composite ABC (total score) is the sum of the raw scores from the main domains. These are transformed in standard scores (m.=100;std.=15). The higher the score, better is the adaptive behavior. Sparrow, S., Balla, D., & Cicchetti, D. (1984). Vineland Adaptative Behaviour Scales: Interview edition, Survey form. Circle Pines, MN: American Guidance Service.
  units on a scale
    VABS_COM_baseline | 68.27 (21.53)
    VABS_DLS_baseline | 77.53 (14.05)
    VABS_SOC_baseline | 65.80 (16.79)
    VABS_ABC_baseline | 65.73 (15.56)

OUTCOME MEASURES:

1. Primary Outcome: JAAT_NoFace
Description: Number of fixations on the target object of the joint attention animation of an avatar after the animation starts (e.g. looking at, pointing at) in the Joint-attention assesment task - JAAT_NoFace with no previous fixation on avatar face.. We will use a new task/realistic game that will challenge the detection of initiation of joint attention cues (from avatars - gaze or pointing). The number of correct responses (to particular objects and not to non-object parts of the scene) will be recorded. We will also record incorrect responses to non-pointing body gestures.
Time Frame: 16 weeks, and 6 months after intervention
Measure: Mean (Standard Deviation); unit: Correct Fixations
Groups:
- High Functioning ASD Adolescents and Adults: Positive diagnostic results for ASD in:
  * Autism Diagnostic Interview-Revised;
  * Autism Diagnostic Observation Schedule;
  * The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria.
Arm/Group | High Functioning ASD Adolescents and Adults
Number analyzed (Participants) | 15
Correct Fixations
  16 weeks | 13.73 (8.19)
  6 months after intervention | 15.00 (10.02)

2. Primary Outcome: JAAT_Face
Description: Number of fixations on the target object of the joint attention animation of an avatar after the animation starts (e.g. looking at, pointing at) in the Joint-attention assesment task - JAAT_NoFace with previous fixation on avatar face.. We will use a new task/realistic game that will challenge the detection of initiation of joint attention cues (from avatars - gaze or pointing). The number of correct responses (to particular objects and not to non-object parts of the scene) will be recorded. We will also record incorrect responses to non-pointing body gestures.
Time Frame: 16 weeks, and 6 months after intervention
Measure: Mean (Standard Deviation); unit: Correct Fixations
Arm/Group | High Functioning ASD Adolescents and Adults
Number analyzed (Participants) | 15
Correct Fixations
  16 weeks | 7.80 (8.77)
  6 months after intervention | 7.53 (8.11)

3. Secondary Outcome: ATEC - Autism Treatment Evaluation Checklist
Description: Autism Treatment Evaluation Checklist (ATEC) evaluates the effectiveness of autism treatments - a 1-page form designed to be completed by parents or caretakers. It consists of 4 subtests: I. Speech/Language Communication (14 items, min.0-max.28); II. Sociability (20 items, min.0-max.40); III. Sensory/Cognitive Awareness (18 items, min.0-max.36); and IV. Health/Phys./Behavior (25 items, min.0-max.75). Total score (sum) ranges from min.0-max.179.
  The results reported here correspond to the total ATEC score to be used for comparison at a later date. The lower the score, the fewer the problems.
Time Frame: 16 weeks, and Follow-Up (6 months after intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Functioning ASD Adolescents and Adults
Number analyzed (Participants) | 15
score on a scale
  16 weeks | 24.29 (12.90)
  Follow-up (6 months after intervention) | 18.43 (11.77)

4. Secondary Outcome: VABS - Vineland Adaptive Behaviour Scale
Description: The Vineland Adaptive Behaviour Scale (VABS) is a semi-structured interview designed to assess global adaptive functioning, composed by 3 main domains: Communication COM, Daily Living Skills DLS and Socialization SOC. The Adaptive Behaviour Composite ABC (total score) is the sum of the raw scores from the main domains. These are transformed in standard scores (m.=100;std.=15). The higher the score, better is the adaptive behavior. Sparrow, S., Balla, D., & Cicchetti, D. (1984). Vineland Adaptative Behaviour Scales: Interview edition, Survey form. Circle Pines, MN: American Guidance Service.
Time Frame: 16 weeks, and Follow-Up (6 months after intervention)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High Functioning ASD Adolescents and Adults
Number analyzed (Participants) | 15
units on a scale
  VABS_COM_16 weeks | 71.33 (21.62)
  VABS_COM_Follow-up (6 months after intervention) | 73.14 (17.29)
  VABS_DLS_16 weeks | 81.60 (14.46)
  VABS_DLS_Follow-up (6 months after intervention) | 86.29 (14.02)
  VABS_SOC_16 weeks | 67.67 (16.18)
  VABS_SOC_Follow-up (6 months after intervention) | 71.14 (16.11)
  VABS_ABC_16 weeks | 69.00 (15.20)
  VABS_ABC_Follow-up (6 months after intervention) | 72.00 (13.65)

5. Other Pre Specified Outcome: POMS - Profile of Mood States
Time Frame: 16 weeks plus 6 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: HADS - Hospital Anxiety & Depression Scale
Description: 21-item measure of clinical depression
Time Frame: 16 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Debriefing Interview Questionnaire
Description: Covers: strategies; general experience of the process; adverse effects;
Time Frame: 16 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 10 months (from baseline until 6 months follow-up assessment)
Groups:
- High Functioning ASD Adolescents and Adults: The eligible patients for the study should be high functioning ASD adolescents and adults.
  These participants should also meet all the following inclusion criteria and none of the exclusion criteria. All queries about patient eligibility should be directed to Susana Mouga before registration.
  ● Positive diagnostic results for ASD in:
  * Autism Diagnostic Interview-Revised;
  * Autism Diagnostic Observation Schedule;
  * The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria.
Arm/Group | High Functioning ASD Adolescents and Adults
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-02-14): https://cdn.clinicaltrials.gov/large-docs/25/NCT02445625/SAP_000.pdf
  • Study Protocol (2015-06-24): https://cdn.clinicaltrials.gov/large-docs/25/NCT02445625/Prot_001.pdf